CLINICAL TRIAL: NCT05762003
Title: Czech Pharmaco-epidemiological Real World Data Study Focused on Effectiveness of Different Disease Modifying Drugs
Brief Title: Czech Pharmaco-epidemiological Study on Disease Modifying Drugs
Acronym: CPE
Status: Completed | Type: Observational
Sponsor: IMPULS Endowment Fund (Other)
Responsible Party: Sponsor
Other Study IDs: ML41011
Record Dates: First submitted 2023-02-09; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferons; Glatiramer Acetate; teriflunomide; Dimethyl Fumarate; Alemtuzumab; Cladribine; Fingolimod Hydrochloride; ponesimod; Rituximab; ocrelizumab; ofatumumab; Natalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: interferons, glatiramer acetate, teriflunomide, dimethyl fumarate, alemtuzumab, cladribine, fingolimod, ponesimod, rituximab, ocrelizumab, ofatumumab, natalizumab — Administered as part of routine clinical practice.

SUMMARY:
Multiple sclerosis (MS) is a severe autoimmune disease that affects mainly young individuals. It is estimated that there are 17-20,000 affected persons in the Czech Republic.

Currently, MS remains an incurable but treatable disease. As of now, there are many drugs that are able to reduce the inflammatory part of the disease that prevails in its initial phases. The problem is the great variability of the severity of clinical course (from relatively benign to severe malignant courses) and different responses of particular patients to particular drugs. A personalized approach with long life monitoring and adjustment of treatment according to the activity of the disease is essential.

From this point of view registries represent one of the most important source of long term data that is used for evaluation of effectiveness and safety of different drugs in areal life setting.

The objective of this study is to compare effectiveness and safety profile in MS patients treated with a different Disease Modifying Drugs (DMDs) and Ocrelizumab using data from the real clinical practice from the Czech national multiple sclerosis patient registry (ReMuS).

ELIGIBILITY:
Inclusion Criteria:

* Each participant must provide informed consent to registry ReMuS in accordance with local regulations
* The patient is treated by any kind of DMDs
* Confirmed diagnosis of multiple sclerosis

Exclusion Criteria:

* Patient withdrawal of informed consent to registry ReMuS

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from primary patient care and included in patient registry ReMuS.
Sampling Method: Non-Probability Sample
Enrollment: 17478 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness in relapses | 1 year from DMD initiation
  Measurement of annualized relapse rate (ARR) in patients on different DMDs.
Effectiveness EDSS | 1 year from DMD initiation
  Description of disability measured by Expanded Disability Status Scale (EDSS) of values 0 to 10, where 0 represents no neurological disability due to multiple sclerosis (MS), and 10 represents death due to MS. The EDSS is commonly used among clinicians, and described by Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983; 33(11): 1444-1452.

SECONDARY OUTCOMES:
Description of baseline characteristics of patients treated by different DMDs at the time of DMT initiation | Baseline
  Baseline characteristics (age, sex, disease duration, previous treatment, type of MS) of patients treated with different DMDs
Description of termination of different DMDs treatment | Day of DMD termination, assessed up to 15 years
  Number of patients that terminate treatment on particular DMDs

CONTACTS AND LOCATIONS:
Locations (1):
- IMPULS Endowment Fund, Prague, Czechia